CLINICAL TRIAL: NCT03345186
Title: A Structured Nurse Led Patient Management Programme to Improve Outcomes in Gout: A Randomized Controlled Trial
Brief Title: A Nurse Led Patient Management Programme to Improve Outcomes in Gout
Acronym: BONUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Rheuma_gout_11_17
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Gout; Arthritis; Crystal Arthropathy
Keywords: Outcome; Gout
MeSH Terms: conditions — Gout; Arthritis; Crystal Arthropathies | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Interventional group: structured nurse led patient management programm & sc Control group standard of care (sc) alone
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse led plus standard of care (Experimental): Nurse Led Patient Management Programme to Improve Outcomes in Gout and Standard of care for gout patients, including nurse delivered patient education and follow up
  Interventions: Other: nurse led plus standard of care
- Standard of care (No Intervention): Standard of care for gout patients

INTERVENTIONS:
Other: nurse led plus standard of care — structured nurse led patient management programme: Patient education will be done by a specialised nurse and nurse consultations and phone calls will be done.
  Arms: Nurse led plus standard of care

SUMMARY:
This study evaluates the addition of a structured nurse led patient management programme to standard of care in gout patients. Half of the patient will receive the nurse led programme in addition to standard of care and the other half will receive standard of care only.

DETAILED DESCRIPTION:
There is evidence from other chronic diseases that nurse led care in addition to standard of care ameliorates outcomes.

In gout the primary target is the serum uric acid level (SUA). We intend to demonstrate the superiority of a structured nurse led patient management programme over standard of care in a randomized controlled study.

The primary endpoint is the percentage of patients reaching the target SUA level at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of gout according to aspiration of Monosodium urate (MSU) crystals or positive dual energy computer tomography (DECT) or American college of rheumatology (ACR) criteria 2015 fulfilled (1)
* written informed consent
* age >=18 years
* ability and willingness to follow a fixed outpatient programme as judged by the investigator
* indication for urate-lowering therapy (ULT)
* In case of established disease and intercritical gout a SUA level over 360 umol per liter is mandatory.

Exclusion Criteria:

* informed consent not obtained
* age <18 years
* inability or unwillingness to follow a fixed outpatient programme as judged by the investigator
* no definite diagnosis of Gout
* no indication for ULT or contraindications against ULT
* in case of established disease and intercritical gout a SUA level <360 umol per liter is an exclusion criterion
* Pregnant or breastfeeding women can´t participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Serum uric acid level at 6 months Follow-up | 6 months
  percentage of patients who reach the SUA target level of 360 umol/l

SECONDARY OUTCOMES:
Longterm achievement of the target SUA at 12 months | 12 months
  percentage of patients who reach the SUA target level of 360 umol/l

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Daikeler, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neogi T, Jansen TL, Dalbeth N, Fransen J, Schumacher HR, Berendsen D, Brown M, Choi H, Edwards NL, Janssens HJ, Liote F, Naden RP, Nuki G, Ogdie A, Perez-Ruiz F, Saag K, Singh JA, Sundy JS, Tausche AK, Vazquez-Mellado J, Yarows SA, Taylor WJ. 2015 Gout Classification Criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheumatol. 2015 Oct;67(10):2557-68. doi: 10.1002/art.39254. PMID 26352873